CLINICAL TRIAL: NCT06237556
Title: The Effect of Melatonin on Anxiety and Sleep Quality in the Peri-Operative Course of Adults Undergoing Coronary Artery Bypass Graft Surgery: Prospective Randomized Controlled Study
Brief Title: Melatonin on Anxiety and Sleep Quality in Adults Undergoing Coronary Artery Bypass Graft Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed ashraf abdelaziz bayoumi, Assistant lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Ain Shams University, Egypt., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FMASU MD228/2023
Record Dates: First submitted 2024-01-21; First posted 2024-02-01 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Melatonin; Anxiety; Sleep Quality; Coronary Artery Bypass Graft
MeSH Terms: conditions — Anxiety Disorders; Sleep Initiation and Maintenance Disorders | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Patients in the control group will receive placebo.
  Interventions: Other: Placebo
- Melatonin group (Experimental): Three days before the operation patients will receive 5 mg of melatonin (Melatonin, Nature Made, Canada, and USA) one hour before assigned sleep time until the time of discharge from hospital.
  Interventions: Drug: Melatonin 5 MG

INTERVENTIONS:
Other: Placebo — Patients in the control group will receive placebo.
  Arms: Control group
Drug: Melatonin 5 MG — Three days before the operation patients will receive 5 mg of melatonin (Melatonin, Nature Made, Canada, and USA) one hour before assigned sleep time until the time of discharge from hospital.
  Arms: Melatonin group

SUMMARY:
The objective of this study is to evaluate the effect of melatonin on post operative sleeping quality, anxiety, and post-operative opioid requirements in adults post coronary artery bypass graft (CABG) surgery.

DETAILED DESCRIPTION:
Sleep disturbance is common among patients undergoing coronary artery bypass graft (CABG), especially during the first week of the postoperative period. Sleep disorders result in important impacts on morbidity, mortality, and quality of life.

Many factors are thought to be the cause of sleep disturbance in patients who have undergone CABG. These factors include environmental stimuli (e.g. noise and uncomfortable beds), individual characteristics (e.g. primary sleep disorder and comorbid health), nature of cardiac illnesses, and surgical complications (e.g. incisional pain, use of diuretics and resultant nocturia, dyspnea, and difficulty in finding the proper position to sleep).

Furthermore, decreased plasma melatonin concentrations have been documented during surgery and the postsurgical period in patients having undergone CABG.

Melatonin is a neurohormone originating from the amino acid, tryptophan, and is mainly secreted by the pineal gland into the blood stream and the cerebrospinal fluid. It possesses a circadian secretion pattern with a low blood concentration during the day and a high concentration at night.

ELIGIBILITY:
Inclusion Criteria:

* Age from 40-60 years.
* Both sexes.
* Patients undergoing standard on-pump CABG with the same technique by the same surgical team.

Exclusion Criteria:

* Refusal of procedure or participation in the study by patients.
* Patients with known history of allergy to one of study drugs
* Patients taking psychiatric medications, CNS depressants, and hypnotic drugs.
* Patients with neurological disorders stroke, intracranial hemorrhage and surgery.
* Patients with a history of suffering from any sleep disorder.
* Severe circulatory or respiratory disease.
* Patients with obstructive sleep apnea.
* Cognitive or psychiatric illness that leads to inability to cooperate, speak or provide informed consent

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Quality of sleep | Five days postoperative
  Sleep quality will be evaluated using the Groningen Sleep Quality Score (GSQS), The GSQS consists of 15 questions about the previous night's sleep, answered with Yes or No.

SECONDARY OUTCOMES:
Anxiety | 24 hours postoperative
  The Hamilton Anxiety Rating Scale (HAM-A) is a psychological questionnaire employed by clinicians to rate the severity of anxiety. This scale includes 14 items. Each consists of a number of symptoms, and the symptoms are graded on a scale of zero to four.
  Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Opioid requirements | 24 hours postoperative
  Postoperative analgesia in the ICU was carried out for both groups. All patients received IV fentanyl infusion (0.5ugm/kg/hr) with 15ug bouls if sudden rise in Heart rate or mean arterial blood pressure > 20% of base line to be stopped before extubation, after extubation Paracetamol 1gm was given every 8 hours for all patients, diclofenac 75mg /12hr.
The degree of pain | 24 hours postoperative
  The degree of pain will be assessed using numerical rating scale (NRS) requires for sternal pain, the patient to rate their pain on a defined scale from 0-10 where 0 is no pain and 10 is the worst pain) measured at time intervals: 30 minutes, 6hours, 12hours, and 24h after extubation. If NRS > 4 rescue analgesia will be given in form of IV morphine0.05mg /kg.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.